CLINICAL TRIAL: NCT05756452
Title: Linking Cardiac Autonomic Dysfunction and InfLammation in Patients With Acute Coronary Syndromes: a Complex Puzzle to be Solved With Potential Therapeutic Implications (CADILACS Study)
Brief Title: Linking Cardiac Autonomic Dysfunction and InfLammation in Patients With Acute Coronary Syndromes
Acronym: CADILACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Lanza Gaetano Antonio, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5480
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Acute Coronary Syndrome; Myocardial Ischemia
Keywords: Subclinical inflammation; Autonomic nervous system; Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia; Angina, Unstable | interventions — Immunologic Memory; Physical Examination

STUDY DESIGN:
Intervention Model Description: Investigators will enroll partecipants who have had an acute coronary syndrome (3 months ± 15 days before enrollment) followed up at the Cardiology Unit of the participating centers.
  Based on the coronary angiography results, partecipants will be divided into two groups:
  1. patients with ACS and obstructive CAD;
  2. patients with ACS without CAD, in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partecipants with ACS and obstructive CAD (Experimental): The study is to identify a difference in the correlation between HRV and CRP parameters in ACS patients with or without obstructive CAD
  Interventions: Diagnostic Test: Anamnesis and clinical evaluation
- Partecipants with ACS without CAD, in a 1:1 ratio (Experimental): Evaluate whether cardiac autonomic dysfunction is associated with low-grade systemic inflammation, inflammasome-dependent activation of IL-18 and IL-1β, and Th1/Treg frequency, in patients with ACS with or without obstructive CAD on angiography
  Interventions: Diagnostic Test: Anamnesis and clinical evaluation

INTERVENTIONS:
Diagnostic Test: Anamnesis and clinical evaluation — All partecipants will undergo a global echocardiographic evaluation, a 24-hour ECG Holter recording to assess HRV and blood samples collection for neurotransmitter measurements, platelet activation and reactivity evaluation and inflammatory profile assessment by proteomics analysis, inflammasome activity evaluation, NLRP3, pro-IL-18 and pro-IL-1β expression level by qPCR and epigenetic analysis.
  Other Names: Transthoracic Doppler Echocardiography (TTDE);; 24-hour Holter ECG recording;; Peripheral venous blood sampling

SUMMARY:
Subclinical inflammation plays a critical role in all stages of the atherosclerotic process, from the initiation of the fatty streaks to the development of plaque instability and rupture, causing myocardial ischemia and acute coronary syndromes (ACS).

A few studies have suggested that the autonomic nervous system (ANS) and the inflammatory response are intimately linked. Accordingly, a relation between impaired cardiac autonomic tone and increased markers of inflammation has been reported in healthy subjects as well as in patients with type 1 diabetes mellitus, chronic coronary syndrome or decompensated heart failure.

To get insight in the controversial relationship between cardiac autonomic dysfunction and inflammation in patients with ACS both with and without obstructive CAD and assess the precise mechanisms and molecular pathways by which these two pathophysiological conditions mutually influence each other, to characterize their prognostic implications and identify possible targets for novel therapeutic strategies.

DETAILED DESCRIPTION:
A comprehensive assessment of cardiac autonomic function and inflammatory profile will be performed in ACS patients with obstructive CAD (n=45) or with NO-CAD (n=45) at coronary angiography. In the sub-acute phase (1 to 6 months after the ACS) all patients will undergo a global echocardiographic evaluation, a 24-hour ECG Holter recording to assess HRV and blood samples collection for neurotransmitter measurements, platelet activation and reactivity evaluation and inflammatory profile assessment by proteomics analysis, inflammasome activity evaluation, NLRP3, pro-IL-18 and pro-IL-1β expression level by qPCR and epigenetic analysis. A follow-up to establish clinical conditions of patients will be done after 12 months by direct clinical visit, trans-thoracic echocardiogram to evaluate cardiac remodeling, HRV assessment by 24-hour ECG Holter recording and blood sample collection to evaluate the inflammatory profile as it was assessed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Evidence of previous complete percutaneous revascularization;
* ACS, with or without CAD, experienced in the previous 3 months ±15 days;
* Signed written informed consent.

Exclusion Criteria:

* History of previous acute myocardial infarction (AMI);
* Prior surgical myocardial revascularization via coronary artery bypass graft (CABG);
* Previous incomplete percutaneous myocardial revascularization, as indicated by documentation of residual stenosis >50% or FFR ≤0.8 in any epicardial vessel;
* Killip class III-IV in admission;
* Established cardiovascular disease (assessed by clinical evaluation, physical exam, 12-lead ECG, or transthoracic echocardiogram), such as congenital heart disease, cardiomyopathy, and severe valvular heart disease;
* Serious medical conditions, including severe renal insufficiency (eGFR > 30 ml/min), hepatic insufficiency or cirrhosis, malignancies, COPD (GOLD stage III-IV), and acute or chronic inflammatory diseases;
* Refusal to sign the written informed consent to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between HRV and CRP parameters in ACS patients with obstructive CAD | 12 months
  The primary endpoint of the study is to identify a difference in the correlation between HRV and CRP parameters in ACS patients with or without obstructive CAD.
  This study will be performed through a detailed history and clinical evaluation based on transthoracic Doppler echocardiography (TTDE) and 24-hour Holter ECG recording.
The correlation between HRV and CRP parameters in ACS patients without obstructive CAD | 12 months
  The study is important to identify the differences between HRV and CRP parameters ACS patients without obtructive CAD.
  It is important to group several exams: sample blood, transthoracic Doppler echocardiography (TTDE) and 24-hour Holter ECG recording.

SECONDARY OUTCOMES:
Evaluate cardiac autonomic dysfunction associated to a systemic inflammation | 12 months
  To evaluate whether cardiac autonomic dysfunction is associated with low-grade systemic inflammation, inflammasome-dependent activation of IL-18 and IL-1β, and Th1/Treg frequency, in patients with ACS with or without obstructive CAD on angiography;To evaluate the precise mechanisms and molecular pathways through which cardiac autonomic dysfunction and inflammation influence each other, in order to identify possible targets for new therapeutic strategies;

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS di Roma, Rome, Lazio, Italy